CLINICAL TRIAL: NCT03442062
Title: Impact of AFIX and Physician-to-Physician Engagement on HPV Vaccination in Primary Care: A Randomized Controlled Trial
Brief Title: Quality Improvement Strategies to Increase Human Papillomavirus (HPV) Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); New York State Department of Health (Other Government); Wisconsin Department of Health and Family Services (Other Government); Arizona Department of Health Services (Other Government); Association of Immunization Managers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0146a; 1U01IP001073-01 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Human Papillomavirus Infection
Keywords: quality improvement; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AFIX (Experimental): Clinics randomly assigned to this arm will receive an Assessment Feedback Incentives and eXchange (AFIX) consultation delivered in-person by a state health department immunization specialist.This arm includes ~ 90 high-volume primary care clinics in three states (New York, Wisconsin, Arizona).
  Interventions: Other: Assessment Feedback Incentives and eXchange
- Physician-to-physician engagement (Experimental): Clinics randomly assigned to this arm will receive physician-to-physician (P2P) consultations delivered remotely to providers by physician educators. This arm includes ~90 high-volume primary care clinics in three states (New York, Wisconsin, Arizona).
  Interventions: Other: Physician-to-physician engagement
- AFIX + P2P (Experimental): Clinics randomly assigned to this arm will receive both an Assessment Feedback Incentives and eXchange (AFIX) consultation and a physician-to-physician (P2P) consultation.This arm includes ~90 high-volume primary care clinics in three states (New York, Wisconsin, Arizona).
  Interventions: Other: Assessment Feedback Incentives and eXchange; Other: Physician-to-physician engagement
- Active Intervention Control (Other): Clinics randomly assigned to this arm will receive a brief non-HPV vaccine related quality improvement consultation. This arm includes ~90 high-volume primary care clinics in three states (New York, Wisconsin, Arizona).
  Interventions: Other: Active Intervention Control

INTERVENTIONS:
Other: Assessment Feedback Incentives and eXchange — The adolescent AFIX (Assessment, Feedback, Incentives, and eXchange) Program is a quality improvement strategy developed by the CDC to improve the immunization practices and vaccination coverage levels of public and private health care providers. It has four main components: 1) Assessment of a provider's current immunization practices and vaccination levels, 2) Feedback of the assessment results and strategies to improve coverage levels, 3) Incentives to improve coverage levels, and 4) eXchange of information and resources necessary to facilitate improvement. Relevant AFIX information will be communicated to vaccine providers using several intervention and quality improvement components.
  Other Names: AFIX
  Arms: AFIX; AFIX + P2P
Other: Physician-to-physician engagement — Physician-to-physician engagement is a quality improvement strategy in which trained physician educators deliver a 60 minute consultation via interactive webinar. The consultations will be delivered to providers in primary care clinics and will include didactic instruction on HPV-related cancers, HPV vaccination, communication training, and assessment and feedback about each clinics' vaccination coverage.
  Other Names: P2P
  Arms: AFIX + P2P; Physician-to-physician engagement
Other: Active Intervention Control — Active Intervention Control will be a remotely delivered quality improvement strategy on a clinical topic other than HPV vaccination.
  Other Names: Control
  Arms: Active Intervention Control

SUMMARY:
HPV vaccination is at lower levels than the national goals. This study will evaluate the effectiveness of quality improvement strategies for increasing HPV vaccination coverage among adolescents in primary care clinics.

DETAILED DESCRIPTION:
The University of North Carolina will test the effectiveness of the Center for Disease Control and Prevention's AFIX model, physician-to-physician engagement, and both strategies in combination, for increasing HPV vaccination coverage among adolescents in primary care clinics. AFIX (Assessment, Feedback, Incentives and eXchange) consists of brief quality improvement consultations that immunization specialists from state health departments deliver to vaccine providers in primary care settings. Using immunization registry data, the specialist evaluates the clinic's vaccination coverage and delivers education on best practices to improve coverage. Physician-to-physician (P2P) engagement consists of physician educators providing feedback about clinics' current HPV vaccination coverage and in-depth training about how to make strong and effective HPV vaccination recommendations to primary care providers via remote webinar consultations. Physician educators will also use immunization registry data to provide feedback on clinics' vaccine coverage. The investigators will compare changes in HPV vaccination coverage before and after intervention for high-volume primary care clinics in four study conditions: AFIX consultations delivered in-person by state health department immunization specialists (AFIX group), physician-to-physician consultations delivered remotely by trained physician educators (P2P group), both AFIX and P2P consultations in combination (AFIX + P2P group), or no HPV quality improvement intervention (control group). In each state, 30 clinics will be randomly assigned to each study arm, for a total of 120 clinics per state, or 360 clinics overall. As a secondary endpoint, we proposed to evaluate the impact of intervention "booster" visits delivered at 12-months post-intervention. However, the CDC has recently changed the AFIX program so that the desired comparison is no longer possible. Therefore, we have eliminated booster visits. This change does not affect our primary endpoint. The primary objective of this study is to compare the change in coverage for HPV vaccine initiation among 11-12 year old patients, from baseline to 12-month follow-up. Secondarily, the study will compare the change in coverage for other vaccines, age groups and time periods.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric or family medicine clinics or practices in New York, Wisconsin, or Arizona with at least 200 active records for patients, ages 11-17, in their states' immunization information systems.

Exclusion Criteria:

* Less than 200 active records for patients between 11-17

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds at 12 months | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12- year old patients, as measured by states' immunization information system (IIS) records

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds at 6 months | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (≥1 dose), 11-12 year olds at six months by state | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI or AZ)
HPV vaccination (≥1 dose), 11-12 year olds at 12 months by state | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI or AZ)
HPV vaccination (≥1 dose), 11-12 year olds at 18 months | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (≥1 dose), 11-12 year olds at 18 months by state | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI, or AZ).
HPV vaccination (completion according to the Advisory Committee on Immunization Practices (ACIP) guidelines), 11-12 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 11-12 year olds at six months by state | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI, or AZ)
HPV vaccination (completion according to ACIP guidelines), 11-12 year olds at 12 months | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 11-12 year olds at 12 months by state | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI, or AZ)
HPV vaccination (completion according to ACIP guidelines), 11-12 year olds at 18 months | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 11-12 year olds at 18 months by state | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY, WI, AZ)
HPV vaccination (≥1 dose), 13-17 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (≥1 dose), 13-17 year olds at 12 months | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (≥1 dose), 13-17 year olds at 18 months | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine initiation (≥1 dose), among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 13-17 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 13-17 year olds at 12 months | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion, among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 13-17 year olds at 18 months | Eighteen months
  Coverage change from baseline to eighteen months in HPV vaccine completion, among 13- to 17- year-old patients, as measured by states' IIS records

OTHER OUTCOMES:
Tetanus, diphtheria, and acellular pertussis (Tdap) vaccination, 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in Tdap vaccination among 11- to 12-year-old patients, as measured by states' IIS records
Meningococcal vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in meningococcal vaccination (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina; Melissa B Gilkey, PhD, Principal Investigator — University of North Carolina
Locations (3):
- United States (3):
  - Arizona Department of Health Services, Phoenix, Arizona
  - New York State Department of Health, Albany, New York
  - Wisconsin Department of Health Services, Madison, Wisconsin